CLINICAL TRIAL: NCT03507426
Title: Retrobulbar Block Versus Ketamine Infusion as Adjuvants to General Anesthesia for Post-operative Pain Control After Enucleation
Brief Title: Retrobulbar Block Versus Ketamine Infusion for Post-enucleation Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nazmy Edward Seif (Other)
Responsible Party: Sponsor-Investigator, Nazmy Edward Seif, Clinical Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RBKIPEA
Record Dates: First submitted 2018-04-15; First posted 2018-04-25 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Enucleated; Eye; Evisceration; Operation Wound; Pain, Postoperative
Keywords: Retrobulbar block; Ketamine; Ocular enucleation; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Ketamine; Analgesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Retrobulbar group (Active Comparator): Retrobulbar block
  Interventions: Procedure: Retrobulbar block
- Ketamine group (Active Comparator): Intravenous analgesia
  Interventions: Procedure: Ketamine
- Control group (No Intervention): General anesthesia alone

INTERVENTIONS:
Procedure: Retrobulbar block — Patients will receive a single retrobulbar injection with 3-4ml of an equal mixture of Lidocaine 2% & Bupivacaine 0.5% + Hyaluronidase (10 IU/ml), after induction of general anesthesia.
  Other Names: Local analgesia
  Arms: Retrobulbar group
Procedure: Ketamine — Patients will receive a 0.5 mg/kg bolus followed by an infusion of 0.25 mg/kg/h of intravenous Ketamine, after induction of general anesthesia.
  Other Names: IV analgesia
  Arms: Ketamine group

SUMMARY:
This study compares the efficacy and safety of two techniques, retrobulbar block versus intra-operative ketamine infusion, for control of post-operative pain occurring in patients undergoing ocular enucleation or evisceration performed under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Ocular enucleation candidate patients
* Ocular evisceration candidate patients

Exclusion Criteria:

* Any condition contra-indicating general or local anesthesia
* Allergy to any of the drugs used during the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Time to the first post-operative rescue analgesia. | 24 hours
  Time (measured in minutes) elapsed till the patient requires to receive his first post-operative rescue analgesic dose.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M El-Badawy, MD, Study Chair — Kasr Al-Ainy Hospital, Cairo University; Nazmy E Seif, MD, Study Director — Kasr Al-Ainy Hospital, Cairo University
Locations (1):
- Kasr Al-Ainy Hospital, Cairo University, Cairo, Egypt